CLINICAL TRIAL: NCT04696965
Title: Appropriate Inhaler Use of Tiotropium As Add-on Therapy to Inhaled Glucocorticoids (ICS) with Long-acting Beta-agonists (LABA) in Adult Patients with Symptomatic Asthma: the Impact of Checking and Correcting Inhaler Technique in Real World
Brief Title: Appropriate Inhaler Use of Tiotropium As Add-on Therapy in Symptomatic Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ting-Yu Lin, Attending physician, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202002047B0
Record Dates: First submitted 2020-12-23; First posted 2021-01-06 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Asthma
Keywords: Tiotropium; Inhaler technique; Asthma
MeSH Terms: conditions — Asthma | interventions — docusate sodium mixt. with phenolphtalein

STUDY DESIGN:
Intervention Model Description: Brief summary of protocol At visit 1, patients characteristics, lung function, cognition function, HRV, CRC and FeNo will be recorded. Randomization by stratification with cognition function will be done but both arms receive usual verbal instruction of inhaler steps.
  At visit 2, inhaler step errors will be recorded 1 months after add-on Tiotropium with ICS+LABA and interventions of education start by correct/recheck strategy in study arm and usual verbal instruction in control arm.
  At visit 3, inhaler step errors will be recorded 3 months after add-on Tiotropium with ICS+LABA as the primary endpoint. Heart rate variability (HRV), cardiopulmonary coupling (CRC) and FeNo will be checked.
  Other endpoints, e.g. lung function, PEFR, exacerbation will be evaluated at V3 and V4 (6 months after V1), V5 (9 months after V1) and V6 (12month after V1)
Who Masked: Participant
Masking Description: The subjects enrolled will be informed the purpose of this study is to evaluate the inhaler step errors after add-on tiotropium with the other ICS+LABA inhaler and how the education improve patients to reduce the error rate. The subjects are not aware the different methods of study arm and control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Correct/recheck strategy (Experimental): Patients of study arm will be asked to show how they use their two inhalers and identify errors using a device-specific checklist by research assistant. Research assistant then show the patient how to use these devices correctly and give the checklist including the steps patients did wrong. After teaching by the research assistant, patients were asked to demonstrate the correct way of wrong step(s) they made at beginning.
  Interventions: Other: Correct/recheck strategy
- Usual verbal instruction (Active Comparator): Patients of control arm will be asked to show how thy use their two inhalers and identify errors using specific check list by research assistant. The educational nurse will give verbal instruction.
  Interventions: Other: Usual verbal instruction

INTERVENTIONS:
Other: Correct/recheck strategy — One month after recruitment and every 3 months. 1. Check the inhaler step errors of patients by research assistant; 2.Demonstrate the right way by research assistant; 3. give the inhaler check list with marks of the wrong step(s) patients made to patients and 4. confirm the patients do the right way of the previous wrong step(s).
  Arms: Correct/recheck strategy
Other: Usual verbal instruction — One month after recruitment and every 3 months.1. Check the inhaler step errors of patients by research assistant; 2. Verbal instruction with a physical demonstration will be given by educational nurse in usual care.
  Arms: Usual verbal instruction

SUMMARY:
This pragmatic, two-arm, randomized controlled trial study aim to survey the inhaler errors of add-on tiotropium therapy with ICS+LABA in real-world practice of asthma patients and the efficacy of recheck stratage of inhaler skills. Patient characteristics and inflammatory features will be evaluated prospectively for association of asthma control by add-on tiotropium.

DETAILED DESCRIPTION:
1. The clinical efficacy of tiotropium as add-on treatment to ICS with a LABA have been demonstrated in clinical trials in adult patients with symptomatic asthma.
2. Certain patients of daily care, like patients with smoking asthma, late onset asthma or asthma with chronic airway obstruction are often excluded from clinical trials.
3. Studies have shown the cognitive function of patients with COPD is impaired. When mixed types of inhaler devices are prescribed, the multiple steps of different devices may ensure complexity and confusion for patients, which may compromise the efficacy of add-on therapy. The inhaler error of add-on tiotropium treatment in real-world asthma treatment is unknown.
4. The improvement of step errors after varieties of teaching intervention is around 30~50%. Strategy of recheck inhaler technique recommended by the treatment guideline may optimized inhaler use. (https://ginasthma.org/gina-reports/).
5. Factors like responseness of short-acting bronchodilators and cholinergic tone have been reported as predictors of a positive clinical response of add-on tiotropium. However, more specific physiological or inflammatory factors. e.g. exhaled nitric oxide test (FeNo), and para symptomatic function and cardiac-pulmonary interaction have not been evaluated prospectively.
6. This pragmatic, two-arm, randomized controlled trial study aim to survey the inhaler errors of add-on tiotropium therapy with ICS+LABA in real-world practice of asthma patients and the efficacy of recheck stratage of inhaler skills. Patient characteristics and inflammatory features will be evaluated prospectively for association of asthma control by add-on tiotropium.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20 to 75 years old asthmatic patients under regular treatment
2. Received medium to high dose ICS with LABA at least 3 months
3. Persistent asthma related symptoms: asthma control questionnaire (ACQ-7>1.5)
4. Physicians in charged prescribed Tiotropium as add-on therapy according to clinical judgement.

Exclusion Criteria:

1. Refuse to provide inform consent
2. Pregnancy or breastfeeding women
3. Patients with chronic obstructive pulmonary disease
4. Using other Long-acting Muscarinic Antagonists e.g. Sebree, Ultibro, Anoro and Spiolto

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Errors rate of Inhaler steps | 3 months
  The improvement of inhaler steps errors after recheck stratage after 3 month of add-on tiotropium and ICS+LABA

SECONDARY OUTCOMES:
Asthma control | 3 months
  The improvement of asthma control evaluated by Asthma Control Test (ACT). The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
Asthma control | 3 months
  The improvement of asthma control evaluated by Asthma Control Questionnaire-7 (ACQ-7).
  ACQ-7 is 7-point scale (0=no impairment, 6= maximum impairment for symptoms and rescue use; and 7 categories for FEV1%)
Forced expiratory volume in one second (FEV1) before bronchodilation | 3 months
  The improvement of FEV1 before bronchodilation evaluated by spirometry after 3 month of add-on tiotropium and ICS+LABA
Acute exacerbation | 3, 6,9 and 12 month
  The rate of acute exacerbation in one year

OTHER OUTCOMES:
Correlation of the errors rate of Inhaler steps and mini-cog score | 1 month
  The mini-cog score will be evaluated when patient recruitment. The mini-cog is score of five-points in total, a score of zero, one or two indicates a concern in cognitive functioning.
  The error of inhaler steps will be recorded one month after 3 month of add-on tiotropium and ICS+LABA.
  Correlation will be tested via Pearson's test or Sperman rank correlation test.
Correlation of the errors rate of Inhaler steps and poor asthma control | 3 month
  The error of inhaler steps will be recorded one month after add-on tiotropium therapy.
  Asthma control will be evaluated by Asthma Control Test (ACT) 3 months after 3 month of add-on tiotropium and ICS+LABA.
  Correlation will be tested via Pearson's test or Sperman rank correlation test. The distribution of errors rate of inhaler steps between patients with asthma well control (ACT>19) and patients with asthma poor control (ACT<=19) will be tested by Mann-Whitney test.

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Yu Lin, Principal Investigator — Chest department, Chang-Gung Memorial Hospital, Linkou branch
Locations (1):
- Department of Thoracic Medicine, Chang Gung Memorial Hospital, Taoyuan District, Taiwan